CLINICAL TRIAL: NCT01980134
Title: Multicenter, Open, Prospective Study on Modified Resect and DIScard Strategy of Small Colonic Lesions Using WavSTAT4 Optical Biopsy System: The MORDIS Study Clinical Investigational Plan
Brief Title: The MORDIS Study Clinical Investigational Plan
Acronym: MORDIS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: SpectraScience (Other)
Collaborators: Azienda Ospedaliera Universitaria Policlinico (Other); European Institute of Oncology (Other); Institut des Maladies de l'Appareil digestif (Unknown); European Georges Pompidou Hospital (Other); KU Leuven (Other); Innere Medizin I Interdisziplinäre Endoskopie Universitätsklinikum Tübingen (Unknown); University of Erlangen-Nürnberg (Other); Copenhagen University Hospital at Herlev (Other); Skane University Hospital (Other); Institute for Clinical and Experimental Medicine (Other Government)
Responsible Party: Sponsor
Other Study IDs: MORDIS Study 010044-002
Record Dates: First submitted 2013-11-01; First posted 2013-11-08 (Estimated); Last update posted 2016-04-14 (Estimated); Status verified 2016-04

CONDITIONS: Adenoma
Keywords: adenomatous colorectal lesions; colorectal polyps; polyps
MeSH Terms: conditions — Adenoma; Polyps

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Samples will be sent for pathological examination and potentially used for other research purposes.
Oversight: Data Monitoring Committee: No

SUMMARY:
To demonstrate the use of WavSTAT4 system during colonoscopy in identifying diminutive colorectal lesions (e.g. hyperplastic polyps) that can be resected and discarded (or even left in-situ) without adverse clinical impact.

DETAILED DESCRIPTION:
To demonstrate the performance of the WavSTAT4 Optical Biopsy System when used at multiple centers.

Endpoint targets are based on the ASGE PIVI recommendations on real-time endoscopic assessment of the histology of diminutive colorectal polyps.

* Primary endpoint: To demonstrate potential of the WavSTAT4 Optical Biopsy System to predict adenomatous histology with a NPV > = 90% for diminutive colorectal lesions.
* Secondary Endpoint: To show that use of the WavSTAT4 system used to determine histology of colorectal polyps ≤5 mm in size, when combined with the histo- pathologic assessment of polyps >5 mm in size, provides a ≥ 90% agreement in assignment of post-polypectomy surveillance intervals when compared to decisions based on pathology assessment of all identified polyps.

ELIGIBILITY:
Inclusion Criteria:

* Male and Female > 18 years
* Standard indication for colonoscopy OR CRC screening OR follow-up examination after the diagnosis of one or more established polyps OR polypectomy (analysis of polyps other than the intended polypectomy)
* Written informed consent

Exclusion Criteria:

* Inflammatory bowel disease
* Hereditary/genetic polyposis syndromes

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: ~1200 patients ≥ 18 years of age at the time of enrollment showing presence of diminutive colorectal polyps.
Sampling Method: Non-Probability Sample
Enrollment: 1200 (Estimated)
Dates: Start 2013-12; Primary Completion 2016-08 (Estimated); Study Completion 2016-11 (Estimated)

PRIMARY OUTCOMES:
To demonstrate potential of the WavSTAT4 Optical Biopsy System to predict adenomatous histology with a NPV > = 90% for diminutive colorectal lesions. | WavSTAT4 Optical Biopsy System gives real-time result. Outcomes are measured when comparing the physician and WavSTAT4 system result to pathology results, which usually take one to two weeks.
  The WavSTAT4 Optical Biopsy System result will be compared to physician visual diagnosis as well as the subsequent pathological report.

SECONDARY OUTCOMES:
Improved determination of post-polypectomy surveillance intervals | Outcome is measured when patients return for routine follow up. which is a long-term study as patients are not usually requested to return for another colonoscopy for many years.
  To show that use of the WavSTAT4 system used to determine histology of colorectal polyps ≤5 mm in size, when combined with the histo- pathologic assessment of polyps >5 mm in size, provides a ≥ 90% agreement in assignment of post-polypectomy surveillance intervals when compared to decisions based on pathology assessment of all identified polyps.

CONTACTS AND LOCATIONS:
Overall Officials: Guido Costamagna, MD, Principal Investigator — Policlinico Gemeli, Roma, Italy
Locations (6):
- Klinika Hepatogastroenterologie Ikem, Prague, Czech Republic, Czechia
- Herlev Hospital, Herlev, Denmark
- Universitäts Klinikum Tübingen, Tübingen, Germany
- Italy (2):
  - European Institute of Oncology, Milan, Italy
  - Policlinico Universitario Gemeli, Roma, Italy
- SKANE University Hospital, Malmo, Sweden

REFERENCES:
- [Background] Ignjatovic A, East JE, Suzuki N, Vance M, Guenther T, Saunders BP. Optical diagnosis of small colorectal polyps at routine colonoscopy (Detect InSpect ChAracterise Resect and Discard; DISCARD trial): a prospective cohort study. Lancet Oncol. 2009 Dec;10(12):1171-8. doi: 10.1016/S1470-2045(09)70329-8. Epub 2009 Nov 10. PMID 19910250